CLINICAL TRIAL: NCT03428581
Title: Preventing Lymphedema in Patients Undergoing Axillary Lymph Node Dissection Via Axillary Reverse Mapping and Lympho-venous Bypass
Brief Title: Preventing Lymphedema in Axillary Lymph Node Dissection
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James W. Jakub, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-010491; NCI-2022-11065 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-10-23; First posted 2018-02-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Lymphedema; Breast Cancer; Melanoma
Keywords: Axillary; Lymph node; Dissection; Reverse Mapping; Lympho-venous Bypass (LVB); Axillary Reverse Mapping (ARM)
MeSH Terms: conditions — Lymphedema; Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALND with ARM +/- LVB (Experimental): Axillary Lymph Node Dissection (ALND) using Axillary Reverse Mapping (ARM) with Lympho-venous bypass (LVB) will be performed.
  Interventions: Procedure: ALND with ARM +/- LVB
- ALND without ARM +/- LVB (Active Comparator): Axillary Lymph Node Dissection (ALND)
  Interventions: Procedure: ALND

INTERVENTIONS:
Procedure: ALND with ARM +/- LVB — Subjects will undergo removal of the lymph nodes in the underarm or "axilla" area. This is referred to as an axillary lymph node dissection (ALND). The procedure for identifying the drainage of the arm lymphatics during an axillary dissection has been coined axillary reverse mapping (ARM). Lympho-venous bypass (LVB) is a technique incorporated along with the ARM procedure that allows preservation of the lymphatics draining the arm while removing the standard lymph nodes and not compromising the extent of the axillary dissection.
  Arms: ALND with ARM +/- LVB
Procedure: ALND — Prospective and retrospective subjects undergoing an ALND.
  Arms: ALND without ARM +/- LVB

SUMMARY:
The researchers are trying to answer if axillary reverse mapping (ARM) with lympho-venous bypass (LVB) in patients undergoing an axillary lymph node dissection reduces the rate and severity of post-operative lymphedema of the arm.

DETAILED DESCRIPTION:
All subjects will undergo an axillary lymph node dissection (ALND). Cluster randomization will determine which of these subjects will have the ARM with LVB and which subjects will have the ALND without this technique. As a baseline, all subjects will have the circumference of their arms measured and complete a questionnaire about lymphedema. Performing the measurements and answering a questionnaire will be repeated at 6, 12, 24, and 36 months after surgery.

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled to undergo an axillary lymph node dissection
* Patients who in the surgeon's judgement are at high risk to convert to an axillary lymph node dissection based intraoperative findings
* English speaking

Exclusion Criteria

* Prior ipsilateral axillary lymph node dissection
* Prior ipsilateral axillary radiation
* Patients undergoing sentinel lymph node biopsy only or at low risk of converting to an axillary lymph node dissection in the surgeon's judgement
* Previous treatment for lymphedema of either arm or prescribed prophylactic treatment for lymphedema.
* Pregnant patients cannot participate in the substudy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Less than 5% limb volume increase in the study extremity compared to baseline and the control extremity | 36 months following surgery
  Bilateral Limb volume measurements
Less frequently reported symptoms of lymphedema in the study extremity compared to baseline and the control extremity | 36 months following surgery
  Validated patient reported surveys

CONTACTS AND LOCATIONS:
Overall Officials: James W Jakub, MD, Principal Investigator — Mayo Clinic; Mara A. Piltin, DO, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials